CLINICAL TRIAL: NCT03464929
Title: Learning Curves for Airtraq Versus King Vision Laryngoscopes
Status: Completed | Type: Observational
Sponsor: Fundación para la Investigación Biosanitaria del Principado de Asturias (Other)
Collaborators: Hospital Universitario Central de Asturias (Other); Fundación Asturcor (Unknown)
Responsible Party: Sponsor
Other Study IDs: ISPA_CritLab_2
Record Dates: First submitted 2018-03-08; First posted 2018-03-14 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Intubation; Laryngoscopy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Airtraq indirect laryngoscopy: Intubation attempts using Airtraq device.
  Interventions: Device: Airtraq indirect laryngoscopy
- King Vision indirect laryngoscopy: Intubation attempts using King Vision device
  Interventions: Device: King Vision indirect laryngoscopy

INTERVENTIONS:
Device: Airtraq indirect laryngoscopy — Attempt to intubation using the Airtraq device
  Groups: Airtraq indirect laryngoscopy
Device: King Vision indirect laryngoscopy — Attempt to intubation using the King Vision device
  Groups: King Vision indirect laryngoscopy

SUMMARY:
Several videolaryngoscopes have been developed but few have been compared in terms of their learning curves and efficacy. The aim of this study is to compare the learning curves of Airtraq versus King Vision in a group of residents trained in direct laryngoscopy. Four residents will perform, after a short training in manikin, 8 intubations with each device. The sequence of use of the devices will be randomized. Outcome measures will be duration of intubation attempt, glottic visualization and percentage of intubation success.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status classification I-II.
* Elective surgery.
* General anesthesia required.

Exclusion Criteria:

* Bronchoaspiration risk.
* Pharmacological allergies.
* Craniofacial anomalies.
* Body mass index > 30.
* Prior history of airway management complications.
* Presence of clinical signs predictive of difficult intubation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients submitted to elective surgery under general anesthesia.
Sampling Method: Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2018-10-25 (Actual); Study Completion 2019-02-25 (Actual)

PRIMARY OUTCOMES:
Time for intubation | 60 seconds
  Time required from the insertion of the blade beyond the incisors until one complete wave pattern of capnography is monitored.
Glottic visualization | 60 seconds
  Scale of glottic visualization achieved
Intubation success | 60 seconds
  Percentage of intubation success

CONTACTS AND LOCATIONS:
Overall Officials: Félix Ezequiel Fernández-Suárez, MD, Study Director — Hospital Universitario Central de Asturias
Locations (1):
- Hospital Universitario Central de Asturias (HUCA), Oviedo, Principality of Asturias, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Su YC, Chen CC, Lee YK, Lee JY, Lin KJ. Comparison of video laryngoscopes with direct laryngoscopy for tracheal intubation: a meta-analysis of randomised trials. Eur J Anaesthesiol. 2011 Nov;28(11):788-95. doi: 10.1097/EJA.0b013e32834a34f3. PMID 21897263
- [Background] Savoldelli GL, Schiffer E, Abegg C, Baeriswyl V, Clergue F, Waeber JL. Learning curves of the Glidescope, the McGrath and the Airtraq laryngoscopes: a manikin study. Eur J Anaesthesiol. 2009 Jul;26(7):554-8. doi: 10.1097/eja.0b013e3283269ff4. PMID 19522050